CLINICAL TRIAL: NCT02501525
Title: Effect of Ureteral Access Sheath Use on Postoperative Pain Level in Patients Undergoing Retrograde Intrarenal Surgery (RIRS)
Brief Title: Effect of Ureteral Access Sheath Use on Postoperative Pain Level in Patients Undergoing RIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ozcan Kilic, M.D., Assoc. Prof. Dr., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-RIRS-UAS-03
Record Dates: First submitted 2015-07-11; First posted 2015-07-17 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Urolithiasis
Keywords: renal stone; retrograde intrarenal surgery; ureteral access sheath; pain
MeSH Terms: conditions — Urolithiasis; Nephrolithiasis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- UAS (+) (Active Comparator): RIRS with ureteral access sheath: A ureteral access sheath (UAS) will be positioned into the ureter of the patient prior to the insertion of the flexible ureterorenoscope (RIRS).
  Interventions: Device: RIRS with ureteral access sheath
- UAS (-) (Experimental): RIRS without ureteral access sheath: A ureteral access sheath (UAS) will not be positioned into the ureter of the patient prior to the insertion of the flexible ureterorenoscope (RIRS).
  Interventions: Device: RIRS without ureteral access sheath

INTERVENTIONS:
Device: RIRS with ureteral access sheath — Ureteral access sheath will be used during RIRS.
  Arms: UAS (+)
Device: RIRS without ureteral access sheath — Ureteral access sheath will not be used during RIRS.
  Arms: UAS (-)

SUMMARY:
This study will include patients aged between 18 and 70 who will undergo retrograde intrarenal surgery (RIRS) due to renal stone(s). A total of 80 patients (male or female) will be recruited, and will be randomized into 2 groups consisting of 40 patients in each group. The first group of patients will undergo RIRS with a ureteral access sheath (UAS) positioned prior to surgery; and the second group will undergo RIRS without UAS. As use of UAS decreases the pressure in the renal pelvis during RIRS, it is aimed to evaluate whether using UAS or not affects the level of pain felt by patients in the postoperative period.

DETAILED DESCRIPTION:
The level of pain of the patients in both groups will be evaluated by using visual analog score (VAS) and verbal rating score (VRS) in the postoperative 0 min (the moment patients gets consciousness after he/she wakes up from general anesthesia), 10th min, 30th min, 60th min and 120th min.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-70 years old
* Having an indication of retrograde infrarenal surgery (RIRS) due to kidney stone

Exclusion Criteria:

* Patients with uncontrolled diabetes mellitus and diabetic nephropathy
* Patients with blood pressure > 140/80 mmHg despite regular use of antihypertensive agent(s)
* Patients with chronic kidney failure who need dialysis
* Patients who have had prerenal, renal or postrenal acute kidney failure 3 months or much earlier
* Patients who have had pyelonephritis 3 months or much earlier
* Patients younger than 18 years or older than 70 years
* Patients who have undergone a kidney surgery within the last 3 months and have abnormal kidney function tests
* Patients with a concomitant ureter stone who will undergo an endoscopic ureter stone treatment at the same session
* Patients using any kind of medication that can affect his/her perception of pain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Postoperative pain level | Within the first 2 hours after the surgery (RIRS)
  Postoperative pain levels of the patients in both groups will be evaluated by using visual analog score (VAS).
Postoperative pain level | Within the first 2 hours after the surgery (RIRS)
  Postoperative pain levels of the patients in both groups will be evaluated by using verbal rating score (VRS).

CONTACTS AND LOCATIONS:
Overall Officials: Ozcan Kilic, M.D., Principal Investigator — Selcuk University, School of Medicine, Department of Urology
Locations (1):
- Selcuk University, School of Medicine, Department of Urology, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Resorlu B, Unsal A, Gulec H, Oztuna D. A new scoring system for predicting stone-free rate after retrograde intrarenal surgery: the "resorlu-unsal stone score". Urology. 2012 Sep;80(3):512-8. doi: 10.1016/j.urology.2012.02.072. Epub 2012 Jul 26. PMID 22840867
- [Background] Cepeda M, Amon JH, Mainez JA, Rodriguez V, Alonso D, Martinez-Sagarra JM. Flexible ureteroscopy for renal stones. Actas Urol Esp. 2014 Nov;38(9):571-5. doi: 10.1016/j.acuro.2014.03.014. Epub 2014 Jun 2. English, Spanish. PMID 24881777
- [Background] Auge BK, Pietrow PK, Lallas CD, Raj GV, Santa-Cruz RW, Preminger GM. Ureteral access sheath provides protection against elevated renal pressures during routine flexible ureteroscopic stone manipulation. J Endourol. 2004 Feb;18(1):33-6. doi: 10.1089/089277904322836631. PMID 15006050
- [Background] Kourambas J, Byrne RR, Preminger GM. Does a ureteral access sheath facilitate ureteroscopy? J Urol. 2001 Mar;165(3):789-93. PMID 11176469
- [Background] L'esperance JO, Ekeruo WO, Scales CD Jr, Marguet CG, Springhart WP, Maloney ME, Albala DM, Preminger GM. Effect of ureteral access sheath on stone-free rates in patients undergoing ureteroscopic management of renal calculi. Urology. 2005 Aug;66(2):252-5. doi: 10.1016/j.urology.2005.03.019. PMID 16040093
- [Background] Stern JM, Yiee J, Park S. Safety and efficacy of ureteral access sheaths. J Endourol. 2007 Feb;21(2):119-23. doi: 10.1089/end.2007.9997. PMID 17338606
- [Background] Lallas CD, Auge BK, Raj GV, Santa-Cruz R, Madden JF, Preminger GM. Laser Doppler flowmetric determination of ureteral blood flow after ureteral access sheath placement. J Endourol. 2002 Oct;16(8):583-90. doi: 10.1089/089277902320913288. PMID 12470467
- [Background] Torricelli FC, De S, Hinck B, Noble M, Monga M. Flexible ureteroscopy with a ureteral access sheath: when to stent? Urology. 2014 Feb;83(2):278-81. doi: 10.1016/j.urology.2013.10.002. Epub 2013 Nov 12. PMID 24231214